CLINICAL TRIAL: NCT04614532
Title: Recognizing Pain Intensity in Alzheimer's Disease: Autonomic Nervous System Variations and Facial Emotion
Brief Title: Recognizing Pain Intensity in Alzheimer's Disease
Acronym: DOMASNA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reduced recruitment potential for study participants.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20CH158; 2020-A02291-38 (Other: ANSM)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease; Pain; Autonomic Nervous System Disease
Keywords: facial emotion
MeSH Terms: conditions — Alzheimer Disease; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with alzheimer's disease (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: Cold Pressor Test; Other: digital sensor of Nociception Level Index
- control subject (Other): Matching by age (± 5 years), gender, and grade level
  Interventions: Diagnostic Test: cognitive assessment; Other: Cold Pressor Test; Other: digital sensor of Nociception Level Index

INTERVENTIONS:
Diagnostic Test: cognitive assessment — global cognitive assessment :
  * Mini Mental State
  * Evaluation of manual laterality
  * Hospital Anxiety and Depression scale
  * 5 words of Dubois
  * Trail Making Test
  * short battery of the praxies
  * neuropathic pain scale (DN4 in french)
  * Analog Visual Scale for pain
  * Fast Front End Efficiency Battery
Other: Cold Pressor Test — consists of the complete immersion of the participant's arm in a basin of cold water maintained at a temperature.
  The test will be divided into two conditions (pain, no pain). In the first, the container will be filled with cold water. In the second, the water in the container will be at room temperature. The investigators will test each arm. During the immersion of the arm, participants will have to remain silent and remove their arm when the ordeal becomes too painful for the painful condition.
  For the non-painful condition, the immersion time will be determined according to the results of the pre test.
Other: digital sensor of Nociception Level Index — placed on the contralateral index finger with the arm immersed in the tank to measure the variation of physiological parameters.

SUMMARY:
The most common form of dementia is Alzheimer's disease, with 900,000 people affected in France in 2015 and a forecast of 1.3 million in 2020. As a consequence of their advanced age, dementia patients often suffer from pain, mainly musculoskeletal or neuropathic pain. However, the exact prevalence of pain in dementia is underestimated. Indeed, several studies indicate that people suffering from dementia report less pain. This phenomenon is all the more true as the stage of dementia is advanced. In addition, people with dementia receive less pain medication than people without cognitive impairment in similarly painful conditions. Hetero-evaluation alone also seems insufficient, with the result that pain is under-treated compared to patients without cognitive impairment. Better pain screening is a major challenge and self-assessment tools should be favoured as a first line of treatment, even for patients with cognitive impairment. suffering from dementia.

The investigators propose in this work to evaluate the variation of vegetative parameters that accompany a painful stimulus. These variations can be recorded at the cardiac, vascular, pupillary or skin conductance level.

DETAILED DESCRIPTION:
It will therefore be a question of inducing experimental pain in patients with Alzheimer's disease, in the early stages of the disease and to check whether pain-related changes in the autonomic nervous system via the Nociception Level index (NoL® system) differ from a control group of subjects matched in age, gender and education level. To induce pain, the investigators will use the "cold pressor test" technique, which consists of leaving the arm immersed in ice water for as long as the pain is bearable. The investigators will also record before, during and after the immersion, the variations of several parameters derived from the autonomic nervous system during the painful stimulation via the NoL® system. During this experience, the participants will be filmed in their entirety to observe the facial emotions related to pain.

ELIGIBILITY:
Inclusion Criteria for patients with alzheimer's disease :

* Diagnosis of the disease by a hospital doctor after an etiological assessment including at least a cerebral MRI, a neuropsychological assessment and, if possible, dementia markers in the cerebrospinal fluid.
* Mini Mental State Score > 23

Inclusion Criteria for control subject :

- Matching by age (± 5 years), gender, and grade level

Exclusion Criteria for 2 groups :

* presence of pain,
* Presence of mood and/or psychiatric disorders (HAD A ou A scores >7).
* Presence of cardiovascular risk factors and beta-blocker and/or calcium channel blocker therapy.
* Patients under guardianship or curatorship

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Nociception Level Index | 30 minutes
  measured for at least 5 minutes before immersion of the arm to have a control measurement. The measurement will continue throughout the time of immersion of the arm and until the arm is out of the water and returns to the control measurement value. This measurement will be taken via a sensor placed on a finger of the contro-lateral hand.
  an index at 0 = absence of nociception, an index at 100 = maximum nociception

SECONDARY OUTCOMES:
facial recognition | 30 minutes
  The subjects will be fully filmed during the procedure. The video will be analyzed after experimentation, thanks to the Facereader® software. Facereader® is a fully automated system for the recognition of facial expressions, allowing an objective evaluation of the emotion of the topics. It uses the Viola-Jones algorithm allowing a 3D modeling of the face as well as the taking in account of the texture of the face. Then, each unit of action of the Facial Action Coding System (FACS) will be assigned to the face. of the patient. The five facial expressions of pain will be integrated into the software allowing them to be automatic recognition. The parameters used will be the intensity of the emotion expression (from 0 to 100).

CONTACTS AND LOCATIONS:
Overall Officials: Céline BORG, MD, Principal Investigator — CHU of Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No